CLINICAL TRIAL: NCT01699217
Title: Front-line Nilotinib Treatment of BCR-ABL+ Chronic Myeloid Leukaemia in Chronic Phase. An Observational Multicentre Study of the GIMEMA CML WP.
Brief Title: Front-line Nilotinib Treatment of BCR-ABL+ Chronic Myeloid Leukaemia in Chronic Phase
Acronym: CML0912
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: CML0912
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Chronic Phase Philadelphia Positive; BCR-ABL Positive; Chronic Myeloid Leukaemia
Keywords: Chronic Myeloid Leukaemia; Philadelphia positive; BCR-ABL positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The GIMEMA CML Working Party promotes a multicentre, observational, prospective study of CML patients treated frontline with NIL. Patients will be followed for 5 years. This study will help the definition of guidelines for the treatment of CML patients in early CP.

DETAILED DESCRIPTION:
The primary objective of the study is to describe the stability of molecular response with NIL as frontline therapy in newly diagnosed, unselected, CP CML patients, in an independent, investigator-initiated observational study. Imatinib mesylate (IM), a protein tyrosine kinase inhibitor (TKI) targeting BCR-ABL, has become in the last decade the standard of care for Chronic Myeloid Leukaemia (CML) in chronic phase (CP)1,2. Nilotinib (NIL) is a second generation TKI, effective in IM-resistant and IM-intolerant patients, which demonstrated superior efficacy to IM in early CP BCR-ABL+ CML patients3. Currently, the most important target of the treatment of CML with TKIs is the major molecular response (MMR), defined as a ≥ 3 log reduction in BCR-ABL/ABL transcript level, marker of better long-term outcome. With imatinib therapy, achieving a MMR correlates with an improved probability of a durable cytogenetic remission30. Results from IRIS suggest that a MMR after 12 months of imatinib therapy may be a marker of stable response. Further on, the IRIS study showed that patients with a MMR after 12 months of therapy had a significantly better probability of disease-free survival compared with those in complete cytogenetic remission, but not in MMR31. Moreover, obtaining an undetectable BCR-ABL transcript level is extremely relevant in order to consider TKIs discontinuation. This condition is known as "Complete Molecular Response" (CMR) and is further defined according to the sensitivity achieved (for the definition see the "Criteria of evaluation" section). As far as treatment discontinuation, two experiences have been published so far, aimed at evaluating the persistence of the CMR after imatinib discontinuation. The first was a pilot study32 where 12 patients were included. These 12 patients discontinued imatinib after at least 2 years of CMR (median duration of negativity, 32 months). Six patients displayed a molecular relapse with a detectable BCR-ABL transcript at 1, 1, 2, 3, 4, and 5 months. Imatinib was then reintroduced and led to a novel molecular response. Six other patients (50%) still have an undetectable level of BCR-ABL transcript after a median follow-up of 18 months (range, 9-24 months). The results of this pilot trial have been confirmed and extended in a second trial, the STIM trial33: 100 patients were enrolled, median follow-up 17 months, 69 patients with at least 12 months follow-up: 42 (61%) of these 69 patients relapsed (40 before 6 months, one patient at month 7, and one at month 19). At 12 months, the probability of persistent CMR for these 69 patients was 41% (95% CI 29-52). All patients who relapsed responded to reintroduction of imatinib. An increase of the CMR rate could possibly translate in a higher proportion of patients candidate to stopping anti-CML treatment, with higher probability of remaining disease-free in the long term. The advantages of this possible future scenario could be: first, the possibility of treatment discontinuation at least in patients with chronic clinical adverse events; second, a potential reduction of the costs of TKI treatment (after the introduction of TKI, the costs of CML treatment is increasing year by year, with the increasing prevalence of CML patients). Standardized molecular monitoring has become widely available in Europe through the efforts of EUTOS cooperation19 and now allows for the generation of comparable data on the residual disease using recalculation on the international scale despite these data being analyzed in many different laboratories. These advances in the standardization of molecular responses and the improvement of targeted therapy have allowed for comparable response assessment across Italian Centres and early treatment optimization of patients.

In summary, 1) monitoring of molecular response and of deep and sustained molecular response, provides a straightforward opportunity to assess patients' response and possible prognosis in the use of targeted therapy. 2) Most data on second generation TKIs are from company-sponsored studies generally implemented in selected referral centres. 3) The detailed description of the kinetic of the molecular response and, particularly, the rate of stable MR4, potentially related in turn with a subsequent treatment discontinuation, within the frame of a long-term post-marketing surveillance observational trial offered to all eligible patients followed at a nation-wide, independent multicentre group is the core distinctive feature of this observational trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: >=18 years;
* Patients with chronic phase Ph+ and/or BCR-ABL+ CML, newly diagnosed (less than 6 months);
* Prior treatment with Hydroxyurea or Anagrelide is allowed;
* Prior treatment with IM for less than 30 days is allowed;
* Signed written informed const according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

* Patients who are pregnant (negative pregnancy test is requested within 2 days before nilotinib start) or breast feeding, or adults of reproductive potential not employing an effective method of birth control.
* Newly diagnosed Ph+ and/or BCR-ABL+ CML patients in advanced phases (accelerated or blastic phase).
* Prior treatment with nilotinib, dasatinib, or other tyrosine-kinase inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment decision is at the discretion of the investigator and must not be made on the basis of this observational study. Patients should have their treatment initiated in accordance with the summary of product characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2013-06-21 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
The rate of confirmed MR4 | At 24 months from study entry

SECONDARY OUTCOMES:
The rate of MMR | At 24, 36, 48, and 60 months from study entry.
The rate of MR4 | At 24, 36, 48, and 60 months from study entry.
The rate of MR4.5 | At 24, 36, 48, and 60 months from study entry.
The rate of confirmed MR4 | At 36, 48, and 60 months from study entry.
The rate of stable MR4 | At 24, 36, 48, and 60 months from study entry
  (at least three PCR results with MR4 within the last year [± 2 months] and no results > 0.01% during the same period).
The rate of stable MR4.5 | At 24, 36, 48, and 60 months from study entry
  (at least three PCR results with MR4.5 within the last year [± 2 months] and no results > 0.0032% during the same period)
The rate of confirmed loss of MMR (MR3) | At 60 months from study entry
The rate of confirmed loss of MMR | At one year from study entry
The rate of Complete Cytogenetic Response | At one year.
The cumulative rate of permanent NIL discontinuation | At 5 years from study entry
  (for failure [defined according to ELN recommendations 2009], intolerance, and death for any reason; not for patients in ≥ MR4 entering clinical trials exploring nilotinib discontinuation)

CONTACTS AND LOCATIONS:
Overall Officials: Gianantonio Rosti, Pr., Principal Investigator — Department of Hematology and Oncological Sciences, S.Orsola-Malpighi Hospital, University of Bologna
Locations (56):
- Italy (56):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Nuovo Ospedale "Torrette", Ancona
  - Dipartimento Area Medica - Presidio Ospedaliero "C. e G.Mazzoni", Ascoli Piceno
  - Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Policlinico Sant'Orsola Malpighi, Bologna
  - USD Trapianti di midollo per adulti - Cattedra di Ematologia - Università degli Studi di Brescia, Brescia
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - U.O.C. di Onco-Ematologia - Centro di Ricerca e Formazione ad Alta tecnologia nelle Scienze Biomediche, Campobasso
  - US Dipartimentale - Centro per le malattie del sangue - Ospedale Civile - S.Giacomo, Castelfranco Veneto
  - ezione di Ematologia C.T.M.O. Istituti Ospitalieri, Cremona
  - Ospedale Santa Croce Divisione di Ematologia Cuneo, Cuneo
  - Policlinico di Careggi, Università delgi studi di Firenze, Florence
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Clinica Ematologica - DiMI - Università degli Studi di Genova, Genova
  - IRCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - SOC Ematologia e Centro Trasfusionale Ospedale di Ivrea - ASL TO4, Ivrea
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - UO Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale San Gennaro - ASL Napoli 1, Napoli
  - Sez. di Ematologia Clinica Ospedale San Francesco, Nuoro
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2 Prof. Giuseppe Saglio, Orbassano
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - La Maddalena Casa di Cura di Alta Specialità Dipartimento Oncologico di III Livello, Palermo
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - U.O. di Ematologia - Centro Oncologico Basilicata, Rionero in Vulture
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Pronto Soccorso e Accettazione Ematologica - Dipartimento Biotecnologie Cellulari ed Ematologia - Università degli Studi di Roma "Sapienza", Roma
  - Segreteria di Ematologia - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Azienda Sanitaria Locale Viterbo - Polo Ospedaliero Centrale - Ospedale Di Ronciglione - U.O. di Ematologia, Ronciglione
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - SS.C. di Oncoematologia - Dipartimento di Medicina Clinica e Sperimentale - Azienda Ospedaliera - S. Maria Di Terni, Terni
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Sezione di Ematologia - Med.II Div. Presidio Ospedaliero S. Chiara di Trento, Trento
  - Azienda U.L.S.S.9 - U.O. di Ematologia, Treviso
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No